CLINICAL TRIAL: NCT00816543
Title: A Single Arm Phase II Feasibility Study of Neoadjuvant Docetaxel, Oxaliplatin and S-1 Chemotherapy in Potentially Operable Gastric or Gastroesophageal Adenocarcinoma.
Brief Title: Docetaxel + Oxaliplatin + S-1 in Potentially Operable Gastric or Gastroesophageal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_R_03761
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; S 1 (combination); Oxaliplatin

ARMS (1):
- 1 (Experimental): 3 cycles of neoadjuvant chemotherapy of Docetaxel, Oxaliplatin and S-1. Surgery 5 to 6 weeks after completion of the chemotherapy.
  Interventions: Drug: DOCETAXEL; Drug: S-1; Drug: OXALIPLATIN

INTERVENTIONS:
Drug: DOCETAXEL — 50 mg/m² IV as a 1 hour infusion on day 1 for each period of 3 weeks for 3 cycles.
Drug: S-1 — 80mg/m² day 1-14 every 3 weeks for 3 cycles. The curative resection group will receive two oral doses of 40 mg/m²/day for 4 weeks, followed by 2 weeks rest, for 1 year.
Drug: OXALIPLATIN — 100 mg/m² on day 1 as a two-hour IV infusion for each period of 3 weeks for 3 cycles.

SUMMARY:
The primary objective of this trial is:

* To determine whether it is feasible in locally advanced gastric or gastroesophageal cancer to administer 3 cycles of Docetaxel, Oxaliplatin and S-1 as a chemotherapy scheme and also to determine what toxicities are involved.

The secondary objective of this trial are to describe:

* The disease free survival at one and two years in that subgroup of patients that has undergone a R0 resection.
* The downstaging after 3 cycles of chemotherapy, pCR in that subgroup of patients that have undergone an R0 resection and progression-free survival and overall survival at one and two years.

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically confirmed, newly diagnosed, localized gastric or gastro-esophageal adenocarcinoma, that is considered operable.

  * The bulk of disease must be localized in the stomach, although the gastroesophageal junction may be involved.
  * Patients with T3 or T4 carcinoma without (N0) and T2 or T3 or T4 with regional lymph node involvement assessed by EUS, no peritoneal seeding suspected on abdomen-pelvic CT or confirmed by laparoscopy.
* Performance status 0-1 in ECOG scale
* Adequate haematological function and liver and kidney function within 7 days prior to enrollment:

  * Absolute neutrophil count > or = 1.5 x 10^9/L
  * Platelets > or = 100 x 10^9/L
  * Haemoglobin > 10 g/dl
  * Calculated creatinine clearance > or = 60 ml/min
  * Total bilirubin < or = 3 x UNL
  * GOT and GPT < or = 3 x UNL

Exclusion Criteria

* Previous surgery on primary tumour
* Prior palliative surgery (open and closure, passage operation)
* Any other type of tumour (e.g. leiomyosarcoma, lymphoma) or a secondary malignancy, excepting basal cell skin carcinoma or basal cell carcinoma in situ of the cervix which have already been successfully treated
* Distant metastases (M1) including distant nodal Groups (Retropancreatic, para-aortic, portal, retroperitoneal, mesenteric node)
* Any previous palliative, adjuvant or neoadjuvant chemotherapy and/or radiotherapy
* Simultaneous therapy with other anti-tumour drugs
* Ileus, chronic inflammatory intestinal disease or extensive resection of the small intestine and other disorders which limit drug resorption. This includes gastric dumping syndrome, indications of accelerated passage through the small intestine, indications of resorption disorders after intestinal surgery
* Evidence of gastric outlet obstruction and /or severe tumor hemorrhage
* Other anamnestic reaction, serious illness or other medical conditions:

  * Unstable, persistent cardiac disease despite medicinal treatment, myocardial infarction within 6 months before the start of the trial
  * Chronic diarrhoea
  * Neurological or psychological disorders including dementia and seizures
  * Active, non-controllable infection or sepsis
  * Actively disseminated intravascular coagulation
* Symptomatic peripheral neuropathy NCI CTC version 3.0 grade > or = 1
* Hypersensitivity to study drugs
* Patients under anticoagulant therapy with warfarin or other coumarines are excluded from participation.
* Pregnant or lactating (in case of potentially childbearing woman, pregnancy test is positive)
* Patients of child-bearing age or the potential to father a child who refuse to use adequate contraception
* Drug, substance or alcohol abuse

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | At the end of the treatment period

SECONDARY OUTCOMES:
Physical examination | Every 3 months during the study period
Chest X-Ray | Throughout the study period
Computed Tomography scan of the abdomen | Every 6 months during the study period
Gastrofiberscopy | Every 1 year from the completion of the treatment for 2 years
Laboratory analysis | Throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Faith Fung, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Seoul, South Korea